CLINICAL TRIAL: NCT05037058
Title: China Diabetes Cardiovascular Initiative
Acronym: CDCV
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Responsible Party: Principal Investigator, Dong ZHAO, Professor of Beijing Institute of Heart, Lung and Blood Vessel Diseases, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Other Study IDs: CDCV2021
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Quality improvement activities — Quality improvement activities

SUMMARY:
As a collaborative project between American Heart Association, Chinese Society of Cardiology, American Diabetes Association and Chinese Diabetes Society, the China Diabetes Cardiovascular Initiative aims to enhance the attention and awareness of cardiovascular health care professionals (HCPs) in the managements of cardiovascular diseases and diabetes, to reduce diabetes-related complication and minimize adverse events in patients with cardiovascular disease, and to reduce the risk of cardiovascular morbidity and mortality in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized with acute coronary syndrome and diabetes.
2. Aged at least 18 years.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized with acute coronary syndrome and diabetes from 40 tertiary hospitals from China.
Sampling Method: Non-Probability Sample
Enrollment: 9600 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients receiving dual antiplatelet therapy at arrival (within 24 hours) | Duration of hospital stay, an expected average of 1 week
Proportion of STEMI patients receiving fibrinolytic therapy within 30 minutes after arrival among those receiving this treatment | Duration of hospital stay, an expected average of 1 week
Proportion of STEMI patients receiving reperfusion therapy by PCI | Duration of hospital stay, an expected average of 1 week
Proportion of STEMI patients receiving primary PCI within 90 minutes after arrival among those receiving this treatment | Duration of hospital stay, an expected average of 1 week
Proportion of NSTE-ACS patients receiving early cardiac troponin measurement (within 6 hours of arrival) | Duration of hospital stay, an expected average of 1 week
Proportion of NSTE-ACS patients receiving risk stratification at admission | Duration of hospital stay, an expected average of 1 week
Proportion of NSTE-ACS patients receiving PCI within recommended times for patients with high or intermediate risk | Duration of hospital stay, an expected average of 1 week
Proportion of patients prescribed dual antiplatelet medications at discharge | Duration of hospital stay, an expected average of 1 week
Proportion of patients with indications prescribed a beta-blocker at discharge | Duration of hospital stay, an expected average of 1 week
Proportion of patients prescribed a statin at discharge | Duration of hospital stay, an expected average of 1 week
Proportion of patients with indications prescribed an ACE-I or ARB at discharge | Duration of hospital stay, an expected average of 1 week
Proportion of patients that receiving an LDL-C assessment | Duration of hospital stay, an expected average of 1 week
Proportion of patients with evaluation for LV systolic function by echocardiography | Duration of hospital stay, an expected average of 1 week
Proportion of smoking patients that receiving smoking cessation advice/counseling | Duration of hospital stay, an expected average of 1 week
Proportion of patients receiving fasting glucose test at least twice | Duration of hospital stay, an expected average of 1 week
Proportion of patients receiving HbA1C test | Duration of hospital stay, an expected average of 1 week
Proportion of patients prescribed a SGLT-2 inhibitor or a GLP-1 receptor agonist at discharge with cardiovascular disease benefit | Duration of hospital stay, an expected average of 1 week
Proportion of patients with body height and weight measured and documented | Duration of hospital stay, an expected average of 1 week
Proportion of patients receiving guidance on individualized dietary | Duration of hospital stay, an expected average of 1 week
Proportion of patients receiving guidance on individualized physical activity | Duration of hospital stay, an expected average of 1 week